CLINICAL TRIAL: NCT05802186
Title: A Single-Arm Phase II Study of Personalized Dose Guidance for Stereotactic Body Radiotherapy (SBRT) in Patients With Lung Tumors
Brief Title: Stereotactic Body Radiation Therapy Planning With Artificial Intelligence-Directed Dose Recommendation for Treatment of Primary or Metastatic Lung Tumors, RAD-AI Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Varian Medical Systems (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 21L04; NCI-2023-01822 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00217995; NU 21L04 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Lung Carcinoma; Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Lung; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy; X-Rays; Radiosurgery; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (AI-directed analysis, SBRT) (Experimental): Patients undergo radiation planning with AI-directed analysis for dose recommendations with Deep Profiler + iGray software on study. Patients then undergo SBRT on study. Patients also undergo PET, CT, MRI, and/or x-ray imaging during screening and follow-up.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Radiology, Treatment Planning; Radiation: Stereotactic Body Radiation Therapy; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Radiology, Treatment Planning — Undergo radiation planning with AI-directed analysis for dose recommendation
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II trial tests the effectiveness and safety of artificial intelligence (AI) to determine dose recommendation during stereotactic body radiation therapy (SBRT) planning in patients with primary lung cancer or tumors that has spread from another primary site to the lung (metastatic). SBRT uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Even with the high precision of SBRT, disease persistence or reappearance (local recurrence) can still occur, which could be attributed to the radiation dose. AI has been used in other areas of healthcare to automate and improve various aspects of medical science. Because the relationship of dose and local recurrence indicates that dose prescriptions matter, decision support systems to help guide dose based on personalized prediction AI algorithms could better assist providers in prescribing the radiation dose of lung stereotactic body radiation therapy treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To obtain preliminary evidence of efficacy (reduction in local failure free survival) in patients receiving SBRT to the lung with personalized artificial intelligence dose guidance (Deep Profiler + iGray).

SECONDARY OBJECTIVES:

I. To evaluate progression free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) version (v.) 1.1 in patients receiving individualized radiation doses to the lung as recommended by Deep Profiler + iGray.

II. To evaluate respiratory function per the Radiation Therapy Oncology Group (RTOG) Pulmonary Function Scale.

III. To assess toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0 in patients receiving individualized radiation doses to the lung as recommended by Deep Profiler + iGray.

IV. To evaluate the feasibility, defined as 85% receiving within 10% of the projected dose, of implementing the individualized radiation doses recommended by machine learning software (Deep Profiler + iGray) in a clinical practice.

OUTLINE:

Patients undergo radiation planning with AI-directed analysis for dose recommendations with Deep Profiler + iGray software on study. Patients then undergo SBRT on study. Patients also undergo positron emission tomography (PET), computed tomography (CT), magnetic resonance imaging (MRI), and/or x-ray imaging during screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiographic findings consistent with lung cancer or solitary or oligometastatic disease in the lung. Most patients will have primary non-small cell lung cancer. For primary lung cancers, we include lesions with ground glass opacities with a solid component of 50% or greater. Patients with solitary or oligo-metastatic disease in the lung may have any other histology or cancer type
* Patients must have radiographically measurable or evaluable disease per RECIST v. 1.1
* Patients must be age >= 18 years
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients of child-bearing potential (POCBP) must have a negative urine or serum pregnancy test prior to registration on study

  * NOTE: A POCBP is any person with an egg-producing reproductive tract (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Radiation therapy is known to be teratogenic. Patients of child-bearing potential (POCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent, for the duration of study participation, and for 7 days following completion of therapy. Should a patient become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately. People who can impregnate their partners treated or enrolled on this protocol must also agree to use adequate contraception from time of informed consent, for the duration of study participation, and 90 days after completion of administration
* Patients must have the ability to understand and the willingness to sign a written informed consent document. Informed consent must be signed prior to registration on study

Exclusion Criteria:

* Patients who have had prior radiotherapy with radiation field overlap
* For primary lung cancers, patients with ground glass opacities without a solid component will be excluded
* Patients who have not recovered from adverse events confined to the thorax (i.e. pneumonitis, bronchial insufficiency, bronchial hemorrhage, esophagitis) due to prior anticancer therapy (i.e., have residual toxicities >= grade 2) with the exception of alopecia. low blood counts (neutropenia, anemia, etc), or anatomically distinct toxicities (i.e. cystitis)
* Patients who are receiving any other concurrent investigational agents or genotoxic chemotherapy for cancer treatment

  * Note: Patients receiving targeted therapies are permitted to enroll on the study. However, patients must pause treatment with targeted therapy 3 days prior to SBRT and restart medication at least 3 days after SBRT. Concurrent immunotherapy (if not investigational) is permitted. Coronavirus disease 2019 (COVID-19) vaccinations are allowed
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Ongoing or active infection requiring systemic treatment
  * Unstable angina pectoris
  * Stage 3 or greater idiopathic pulmonary fibrosis
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing. Pregnant women are excluded from this study because radiation therapy has teratogenic or abortifacient effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Local failure free survival (LFS) | Assessed at 2 years
  LFS is defined as the length of time after SBRT that the patient survives without local failure (as assessed by tumor imaging).
LFS | Up to 5 years
  LFS data will be collected from the end of SBRT, until the patient experiences recurrence, completes the 5-year follow-up after SBRT, or experiences death from any cause (whichever is sooner).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Assessed at 2 years
  For PFS analysis, disease progression is defined as progressive disease per Response Evaluation Criteria in Solid Tumors version 1.1.
Respiratory function | Up to 30 days
  To assess the respiratory toxicity of SBRT doses as recommended by Deep Profiler +iGray, this endpoint will collect and report the frequency of adverse events by type, severity (grade), timing, and attribution, according the RTOG Pulmonary Function Test Toxicity Scale.
Incidence of adverse events | Up to 30 days
  To assess the Toxicity Profile of SBRT fractions as recommended by Deep Profiler +iGray, this endpoint will collect and report the frequency of adverse events by type, severity (grade), timing, and attribution, according the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0.
Dose recommended | During the 1-2 weeks period of SBRT
  To evaluate if individualized radiation doses recommended by machine learning software (Deep Profiler +iGray) can be implemented in a clinical practice (feasibility), we will assess the adherence of the prescribing physician to the dose recommended by the Deep Profiler +iGray during the 1-2 week period of SBRT. The adherence to the dose recommended by the Deep Profiler +iGray will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Abazeed, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States